CLINICAL TRIAL: NCT05993962
Title: Efficacy of The Daily Consumption of Vitamin B12 Fortified Yoghurt on Vitamin B12 Status of Healthy Older Adults - A Double-blind, Randomized Controlled Trial
Brief Title: Effect of Daily Consumption of Vitamin B12 Fortified Yoghurt on Vitamin B12 Status in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Yvonne Lamers, Associate Professor, Food, Nutrition and Health, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H18-01353
Record Dates: First submitted 2022-12-06; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Vitamin B 12 Deficiency
Keywords: Food fortification; Yogurt; Vitamin B12; Older adults; Fortified food; Yoghurt; Vitamin
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Participants received one daily serving (provided in one cup of 150grams) of unfortified yoghurt for 8 weeks
  Interventions: Other: Control yoghurt
- Fortified group (Experimental): Participants received one daily serving (provided in one cup of 150grams) of yoghurt fortified with vitamin B12 for 8 weeks
  Interventions: Dietary Supplement: Fortified yoghurt

INTERVENTIONS:
Dietary Supplement: Fortified yoghurt — Food-grade vitamin B12 in the form of methylcobalamin (purity: 99%) was used for fortification. Yoghurts were Greek-style and locally produced by a yoghurt company in British Columbia, Canada. The pre-measured vitamin B12 was added into yoghurt vats in amounts that corresponded to the chosen dosage (50 µg of B12 per 150 g). The yoghurt was packaged into white cups, each containing 150 grams of yoghurt, labelled with the date of production and study code.
  Arms: Fortified group
Other: Control yoghurt — Yoghurts were locally produced by a yoghurt company in British Columbia, Canada. Yoghurts produced were Greek-style and packaged into white cups, each containing 150 grams of yoghurt, labelled with the date of production and study code.
  Arms: Control group

SUMMARY:
Older adults are recommended to meet their daily vitamin B12 (B12) requirements by consuming foods with added B12 and/or taking B12 supplements (i.e. sources of free B12) because of an age-related decreased digestion and absorption capacity for food-bound B12. Currently, B12 is not added to foods in Canada, except for simulated dairy and meat products. Yoghurt with added B12 is a novel dairy product that could fill a gap that presently exists in the Canadian market and has the potential to provide Canadian older adults with an alternative dietary source of B12 that could help improve their B12 status. Thus, the objective of this study was to assess the efficacy of the daily consumption of one serving of yoghurt fortified with B12 versus unfortified yoghurt for 8 weeks on the B12 status of healthy older adults, assessed using serum total B12. The primary hypothesis of this study was that the daily consumption of B12-fortified yoghurt would increase serum total B12 concentration of older adults compared to the consumption of unfortified yoghurts.

ELIGIBILITY:
Inclusion Criteria: Non-smoking and apparently healthy female and male volunteers aged 50-75 years, who are comfortable speaking, reading and understanding English.

Exclusion Criteria:

* Chronic health conditions, especially those related to B12 metabolism and the digestive tract. Chronic health conditions include diabetes, cancer, liver disease, psychiatric illnesses (depression, bipolar disorder, schizophrenia, anxiety disorder, eating disorder), cardiovascular disease, renal impairment, pancreatic dysfunction, gastrointestinal diseases (such as, Crohn's disease, Irritable Bowel Syndrome, Colitis, pernicious anemia, Celiac disease, acid indigestion, constipation, diverticulitis/ diverticulosis, gastroesophageal reflux disorder, or atrophic gastritis), total or partial gastrectomy, gastric bypass or other bariatric surgery, ileal resection or organ reconstructive surgery.
* Use of prescription or over-the-counter medications that may interfere with B12 status, i.e., Metformin, anti-cancer treatment, antibiotics, proton pump inhibitors, antacids; the use of high-dose B12 supplements for the last 1 month (e.g., 1000ug of B12 per day); intramuscular B12 injections in the last 1 month; vitamin supplements containing B-vitamins over the past three months; or Brewer's yeast over the past three months.
* Individuals who are unwilling to consume one daily serving of yoghurt for 8 weeks, provide blood samples and measures of height and weight, enroll and start the study in early 2019, or come to the University of British Columbia (UBC) or the BC Children's Hospital Research Institute (BCCHRI) site for study visits.
* Participants with deficient or high serum total B12 concentrations (<148 and >400pmol/L)
* Individuals with allergies or sensitivities to any ingredients of yoghurt (i.e. dairy)
* Individuals who smoke or consume more than one drink containing alcohol each day

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Serum total B12 concentration | Change after 8 weeks of intervention
  Direct biomarker of vitamin B12 status
Serum total B12 concentration | Change after 4 weeks of intervention
  Direct biomarker of vitamin B12 status

SECONDARY OUTCOMES:
Serum holotranscobalamin (holoTC) concentration | Change after 8 weeks
  Direct biomarker of vitamin B12 status
Serum holotranscobalamin (holoTC) concentration | Change after 4 weeks
  Direct biomarker of vitamin B12 status
Plasma methylmalonic acid (MMA) concentration | Change after 8 weeks
  Functional biomarker of vitamin B12 status
Plasma methylmalonic acid (MMA) concentration | Change after 4 weeks
  Functional biomarker of vitamin B12 status
Plasma homocysteine concentration | Change after 8 weeks
  Functional biomarker of vitamin B12 status
Plasma homocysteine concentration | Change after 4 weeks
  Functional biomarker of vitamin B12 status

OTHER OUTCOMES:
Plasma total folate concentration | Change after 8 weeks
  Biomarker for folate status
Plasma total folate concentration | Change after 4 weeks
  Biomarker for folate status

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lamers, PhD, Principal Investigator — Associate Professor, UBC Food, Nutrition and Health
Locations (2):
- Canada (2):
  - BCCHR Clinical Research and Evaluation Unit (CREU), Vancouver, British Columbia
  - UBC Western Nutrition Research Center (WNRC), Vancouver, British Columbia